CLINICAL TRIAL: NCT02099097
Title: Quit IT: Preliminary Testing of a Web-based, 3D Coping Skills Game to Increase Quitting Self-Efficacy for Maintaining Smoking Abstinence Following Hospitalization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: New York University (Other); Muzzy Lane Software (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 14-062
Record Dates: First submitted 2014-03-25; First posted 2014-03-28 (Estimated); Last update posted 2020-12-30 (Actual); Status verified 2020-12

CONDITIONS: Tobacco Use Cessation
Keywords: 3D Coping Skills Game; Quit smoking; 14-062
MeSH Terms: conditions — Tobacco Use Cessation | interventions — Surveys and Questionnaires

ARMS (2):
- Standard Care (Active Comparator): usual care, which consists of four (face-to-face or telephone) counseling sessions with a trained nurse who has expertise in helping cancer patients quit smoking. This is the same as the treatment an MSK patient who enrolls in the MSK smoking cessation program would receive.
  To collect further data to improve the game intervention, the investigators will conduct semi-structured telephone interviews with patients who were randomized to the treatment arm but did not play the game during the one month intervention period. The purpose of the interviews is to elicit qualitative feedback on any barriers that may have prevented participants from playing. At the completion of the intervention period, patients will be asked if they would like to participate in a telephone interview. Telephone interviews will take about twenty minutes and will be held at a time that is convenient for the patient.
  Interventions: Behavioral: Questionnaires; Other: Salvia sample
- Smoking Cues Coping Skills Game (SC+SCCS/Quit IT). (Experimental): Smokers randomly assigned to SC+SCCS/Quit IT will receive all the components of Standard Care. The patient will be oriented and trained face-to-face (during their hospitalization) on use of the game by study staff using an iPad. The orientation and training session will comprise: 1) Overview of the game and its objectives; 2) discussion of the rules of the game; 3) watching a 10 minute tutorial given by the game narrator (avatar); 4) answering all patient questions; and 5) evaluation of the patient's comprehension of game play via a 17 question survey. Once patients have access to QuitIT, they will also receive a set of Coping Cards
  Interventions: Other: web-based video game (Quit IT); Behavioral: Questionnaires; Other: Salvia sample

INTERVENTIONS:
Other: web-based video game (Quit IT)
  Arms: Smoking Cues Coping Skills Game (SC+SCCS/Quit IT).
Behavioral: Questionnaires — In order to maximize survey the response rate, patients will be mailed a reminder letter approximately two weeks before the 1 month follow up surveys are due. If the survey is not returned, patients will be sent additional reminders on the survey due date as well as two weeks past the due date.
Other: Salvia sample — The investigators will inform patients prior to obtaining their self-reports that a saliva test or expired CO sample for those using NRT or electronic cigarettes will be performed to examine recent tobacco exposure.

SUMMARY:
The purpose of this study is to develop and test a web-based game called Quit It that is designed to help smokers who have quit smoking cope with any smoking urges they may have. The purpose of the game is to help people quit and stop people from smoking again.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* English-speaking
* Cancer (solid tumor) diagnosis or mass suspicious of cancer within past six months as per clinical judgment
* Cancer treatment expected plan to include hospitalization for surgical treatment for at least 2 days at MSKCC as per the patients clinical team
* Referred to MSK's Tobacco Cessation Program
* Patient-reported cigarette use within the past 30 days
* Have sufficient sensory acuity (i.e., auditory, visual) and manual dexterity to use a computer game as per judgment of clinician or consenting professional
* Can be reached by telephone

Exclusion Criteria:

* Distant metastatic disease at the time of enrollment
* Major psychiatric illness or cognitive impairment that in the judgment of the investigator would preclude study participation
* Any patients who are unable to comply with the study procedures as determined by the study investigators

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-03-24 (Actual); Primary Completion 2020-12-24 (Actual); Study Completion 2020-12-24 (Actual)

PRIMARY OUTCOMES:
quitting smoking self-efficacy | 1 year
  as measured by the Confidence Questionnaire to assess changes in confidence in being able to resist urges to smoke across everyday situations.

SECONDARY OUTCOMES:
efficacy of the game | 1 year
  on smoking abstinence and relapse prevention. We will examine time to smoking relapse following hospitalization, measured as part of the follow-up Smoking Status 1 month following enrollment. We will also biochemically verify 7-day point prevalence smoking abstinence at the 1 month follow-up assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Jamie Ostroff, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Streck JM, Rigotti NA, Livingstone-Banks J, Tindle HA, Clair C, Munafo MR, Sterling-Maisel C, Hartmann-Boyce J. Interventions for smoking cessation in hospitalised patients. Cochrane Database Syst Rev. 2024 May 21;5(5):CD001837. doi: 10.1002/14651858.CD001837.pub4. PMID 38770804
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/

DOCUMENTS (1):
  • Informed Consent Form (2016-05-19): https://cdn.clinicaltrials.gov/large-docs/97/NCT02099097/ICF_000.pdf